CLINICAL TRIAL: NCT06793345
Title: Moderate Intensity Intermittent Walking Training (MIWT) Improves Thyroid Function and Cardiometabolic Risk Factors in Obese Postmenopausal Women
Brief Title: Walking Training Improves Thyroid and Cardiometabolic Markers in Postmenopausal Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wissal Abassi (Other)
Responsible Party: Sponsor-Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Organization: High Institute of Sports and Physical Education of Kef (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Training and thyroid function
Record Dates: First submitted 2025-01-18; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Hormones; Cardiometabolic Risk Factors
Keywords: Thyroid hormones; Lipid profile; Obesity; Blood pressure; Moderate intensity intermittent walking training; Body composition
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIWT group (Experimental): The MIWT group received moderate intensity intermittent walking training four times per week for 10 weeks.
  Interventions: Other: Moderate intensity intermittent walking training
- Control group (No Intervention): The control group received no intervention for 10 weeks.

INTERVENTIONS:
Other: Moderate intensity intermittent walking training — The intensity of the training is 60 to 80% of 6MWTdistance.
  Arms: MIWT group

SUMMARY:
The goal of this clinical trial is to investigate the impact of a 10-week MIWT program on thyroid hormone levels and key cardiometabolic markers in obese postmenopausal women. The main question it aims to answer is:

Does MIWT enhance thyroid function and reduce cardiometabolic risk factors in this population? Researchers will compare MIWT (designed to MIWT group) to non-training intervention (designed to control group) to see if the training program works to improve thyroid function and cardiometabolic risk factors.

Participants in MIWT group will: perform a 10-week MIWT program, four sessions per week (5 repetitions of 6-min-walking-test (6MWT) at 60-80% of 6MWTdistance measured at baseline, interspersed by 6-min of active recovery between repetitions).

Participants in control group will : not perform any physical training and maintain their usual daily activities.

DETAILED DESCRIPTION:
This study aimed to investigate the impact of a 10-week MIWT program on thyroid hormone levels and key cardiometabolic markers in obese postmenopausal women. Thirty-six obese postmenopausal women (BMI≥30 kg.m-2, aged 50-60 yrs.) were randomized to either a moderate-intensity intermittent walking training (MIWT) group (n=18) or control group (CG, n=18). Participants performed a 10-week MIWT program, four sessions per week (5 repetitions of 6-min-walking-test (6MWT) at 60-80% of 6MWTdistance measured at baseline, interspersed by 6-min of active recovery between repetitions). Body composition, thyroid hormones (thyroid stimulating hormone (TSH) and thyroxine free (FT4)), lipid profile (triglycerides (TRG), total cholesterol(TC), high-density lipoprotein cholesterol(HDLC) and low-density lipoprotein cholesterol(LDLC)), blood pressure (systolic and diastolic blood pressure) and aerobic fitness (6MWT) were determined before and after the MIWT.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index≥ 30 kg.m-2.
* Age between 50 and 60.
* Amenorrhea for >12 months.
* Stable eating habits.

Exclusion Criteria:

* Chronic diseases.
* Medical contraindications to physical activity.
* Hormone replacement therapy.

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-22 (Actual)

PRIMARY OUTCOMES:
Thyroid hormones | At baseline and after ten weeks of MIWT.
  Serum thyroid hormone concentrations are measured from a blood sample (5 ml) obtained from a prominent superficial vein in the antecubital region.
Body composition | At baseline and after ten weeks of MIWT.
  Body composition was assessed using an electronic scale (Tanita BC-533, Tokyo, Japan),
Lipid profile | At baseline and after ten weeks of MIWT.
  Measured by blood samples (5ml) from a prominent superficial vein in the antecubital region.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure | At baseline and after ten weeks of MIWT.
  Systolic and diastolic blood pressure measurements were conducted using an automatic blood pressure monitor (Omron BP652, Omron Healthcare Inc., Vernon Hills, IL, USA).
Heart rate | At baseline and after ten weeks of MIWT
  Heart rate was recorded after 10 minutes of relaxation in a seated position using an automatic blood pressure monitor (Omron BP652, Omron Healthcare Inc., Vernon Hills, IL, USA).
6 min walking test distance | At baseline and after ten weeks of MIWT
  It was recorded using the 6 min walking test.
Perceived exertion rating | At baseline and after ten weeks of MIWT.
  Perceived exertion rating (RPE) was assessed with the extensively validated RPE, a 15-point scale ranging from 6 ("no exertion at all") to 20 ("maximal exertion").

CONTACTS AND LOCATIONS:
Locations (1):
- High Institute of Sports and Physical Education of Kef, Boulifa, Kef Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study are available upon request.